CLINICAL TRIAL: NCT07401498
Title: A Multicenter Prospective Observational Study of the Incidence and Predictors of Complications Directly Related to Lymphadenectomy (LAD) in Surgical Treatment of Non-small Cell Lung Cancer (NSCLC).
Brief Title: Complications Associated With Lymphadenectomy (LAD) in Surgical Treatment of Non-small Cell Lung Cancer (NSCLC).
Acronym: LNDNSCLC-RUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Clinical Oncology Dispensary (Other Government)
Collaborators: National Medical Research Center of Phthisiopulmonology and Infectious Diseases (Other Government); National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6140825
Record Dates: First submitted 2025-12-01; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lymph Node Dissection; Advanced Non-small Cell Lung Cancer (NSCLC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical intervention (Experimental): * Surgical approach: open/VATS.
  * Recorded characteristics: 4L-station dissection (yes/no), recurrent nerve visualization, use of energy devices (specify which: bipolar coagulation, ultrasound, or monopolar energy) on the 4L-station, prophylactic duct clipping (yes/no), number of drains/aspiration mode.
  Interventions: Procedure: Systematic mediastinal nodal dissection (SND); Procedure: Lobe-Specific Lymph Node Dissection (L-SND)

INTERVENTIONS:
Procedure: Systematic mediastinal nodal dissection (SND) — removal of all tissue with lymph nodes in the relevant areas with a minimum of: ≥3 mediastinal stations always including group 7 lymph nodes.
Procedure: Lobe-Specific Lymph Node Dissection (L-SND) — removal of all tissue with lymph nodes in the relevant areas with a minimum of: ≥3 mediastinal stations always including group 7 lymph nodes.

SUMMARY:
Systemic mediastinal lymph node dissection is a standard step in radical surgery for advanced non-small cell lung cancer (NSCLC). However, it does not carry the risks associated with certain procedures (chylothorax, recurrent nerve palsy, diaphragmatic relaxation, intrapleural hemorrhage, injury to other chest organs (esophagus, great vessels), etc.). Data on their incidence and predictors in routine practice are limited.

Objective: To assess trends and characteristics of projects directly related to Lymph Node Dissection and to identify independent risk factors for their development.

DETAILED DESCRIPTION:
Non-small cell lung cancer remains one of the leading causes of cancer-related mortality. Surgical treatment in resectable stages is considered the main radical modality, and systematic mediastinal lymph node dissection is an integral part of this approach. Mediastinal Lymph Node Dissection (MLND) ensures accurate pathomorphological staging, enables detection of subclinical lymph node involvement and improves the quality of locoregional control. At the same time, extending the volume of lymph node dissection increases the invasiveness of the procedure and may lead to serious specific complications.

In routine clinical practice, data on the incidence of these complications and on the risk factors for their development are limited and fragmented, which makes it difficult to assess the risk-benefit ratio when choosing the extent of lymph node dissection for an individual patient.

Published data on the incidence of complications after mediastinal lymph node dissection are highly variable, which is related to differences in study design, complication recording criteria, extent of lymph node dissection and surgeon experience. In addition, most reports are based on data from highly specialized centers and do not fully reflect routine clinical practice. The limited and heterogeneous nature of the available information hinders the development of clear recommendations for risk stratification.

It is assumed that the likelihood of complications is influenced by both surgical factors (extent and anatomical field of lymph node dissection, surgical approach - thoracotomy vs. video-assisted thoracoscopic surgery, duration of the operation, intraoperative blood loss) and patient-related characteristics (age, comorbidities, functional status, tumor location and stage). However, the independent contribution of each of these factors has not been fully defined.

The aim of the present study is to systematize data on the real-world incidence and pattern of complications directly related to Mediastinal Lymph Node Dissection in routine practice and, using multivariable analysis, to identify independent predictors of their development. Evaluating these parameters will make it possible to:

refine the safety profile of mediastinal lymph node dissection;

identify patient groups at increased risk of complications;

optimize the strategy of surgical treatment for advanced non-small cell lung cancer (NSCLC), including the choice of the extent of lymph node dissection and postoperative monitoring.

The findings may serve as a basis for improving clinical guidelines and for a more personalized approach to planning radical procedures in patients with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Clinical stage IA-IIIB NSCLC (TNM 8th edition), oncologically radical resection is planned: anatomical segmentectomy/lobectomy/bilobectomy/pneumonectomy (including sleeve resection).
* LND (systematic) is performed with mandatory inclusion of group 7 (subcarinal) lymph nodes.
* Signed informed consent from all study patients.

Exclusion Criteria:

* Small cell lung cancer, benign and metastatic tumors.
* "Wedge" surgery without any lymph node dissection.
* Nonemergency surgery; conversion is acceptable.
* Patients who cannot complete 30 days of observation (no contact, etc.) should be excluded prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Frequency and outcome after Lymphadenectomy complications within 30 days after surgery | 30 days
  Frequency and outcome after Lymphadenectomy complications within 30 days after surgery (including in-hospital and rehospitalizations): TM&M ≥IIIa.

SECONDARY OUTCOMES:
The frequency of each of the initially obtained complications separately. | 90 days
  Any Lymphadenectomy complications (TM&M I-V), severity profile.
  • Postoperative persistent cough associated with LAE: new or significantly worsened compared to preoperative level; assessment by Visual Analog Scale (VAS) (0-10) and Leicester Cough Questionnaire (LCQ) questionnaire; duration and need for conservative therapy are recorded (initial postoperative assessment at discharge, day 30, day 90).
  Definition of clinically significant cough: ΔVAS ≥2 points or a decrease in the total LCQ score ≥1 point on day 30, after excluding alternative causes (pneumonia, atelectasis, COPD exacerbation, heart failure).
  * Reoperations and invasive interventions for lymphadenectomy complications.
  * Duration of drainage, total hospital stay (days), ICU stay (hours)
  * 30- and 90-day mortality; 30- and 90-day readmission.
  * Voice/dysphagia (Voice Handicap Index questionnaire (short form), if this complication is present), need for medial thyroplasty/injection laryngoplasty at 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Clinical Oncology Dispensary, Ulyanovsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol